CLINICAL TRIAL: NCT07071181
Title: A Randomised, Double-blind Trial to Measure the Effects of Milk-based Drinks on Gut Microbiome, Sleep, and Cardiometabolic Markers in Adults With Poor Sleep
Brief Title: Effects of Milk-based Drinks on Gut Microbiome, Sleep and Cardiometabolic Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Biotiful (Unknown); University of Leeds (Other); Nimble Science Ltd. (Industry)
Responsible Party: Principal Investigator, Tony Lynn, Dr Anthony Lynn, Sheffield Hallam University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: ER72870766; Other (Other Grant/Funding Number: Sheffield Hallam University)
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Sleep; Cardiovascular Diseases; Gut Microbiome; Cognitive Function and Mood; LDL Cholesterol
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Milk

STUDY DESIGN:
Intervention Model Description: This trial conforms to a randomised, double-blind, 2 arm crossover. Participants will consume the active drink or a control drink for 4 weeks before crossing over to the opposite condition after a 4-week washout. Order of drink allocation will be counterbalanced.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Original Kefir (Active Comparator): 250ml of original kefir
  Interventions: Dietary Supplement: Original flavour kefir
- Milk (Sham Comparator): 250 ml of milk
  Interventions: Other: Milk

INTERVENTIONS:
Dietary Supplement: Original flavour kefir — Participants will consume 250ml of original flavour kefir daily for 4 weeks. According to the manufacturer, "packed with billions of live cultures to support Gut health".
  Arms: Original Kefir
Other: Milk — Participants will consume 250 ml milk daily for 4 weeks. This milk will not contain any live cultures.
  Arms: Milk

SUMMARY:
The purpose of this study is to evaluate the effects of kefir on gastrointestinal health, sleep quality, and biochemical parameters in adults who have sleep problems. Further measurements of cognitive function, arterial stiffness and blood pressure will also be assessed.

The following questions will be addressed during the study:

1. What effect does repeated ingestion of kefir have on the gut microbiome and can this positively influence sleep performance (quality and duration) in adults with sleep problems?
2. Does repeated ingestion of kefir impact LDL, triacyglycerols and non-HDLc in adults with sleep problems?
3. What effect does repeated ingestion of kefir have on cognitive function and mood?
4. What effect does repeated ingestion of kefir have on vascular function, inflammation and markers of immunity in adults with sleep problems?

In a randomised, crossover design study, participants will consume 250 ml of kefir (original flavour) or milk for 4 weeks with a 4-week washout.

DETAILED DESCRIPTION:
The gut microbiome is recognized as a key regulator of host health, influencing various physiological processes. Dysbiosis of the gut microbiome has been implicated in a range of adverse health outcomes, including disruptions in sleep architecture and impairments in cardiometabolic function. There is growing interest in identifying dietary interventions that can modulate gut microbiota composition and functionality. In particular, the consumption of fermented foods, such as kefir, has emerged as a potential strategy for promoting microbial homeostasis and improving health outcomes

This study conforms to a randomised, double-blind 2-arm crossover design. Participants will consume either Kefir (original flavour) or milk. Each arm will involve daily consumption of the drink for 4-weeks with a 4 week washout before crossing over to the opposite condition. Drinks will be administered in a counterbalanced order to minimise potential order effects.

The primary outcome of this study is a 5% change in LDL based on a previous study (Bellikci-Koyu et al., 2022).

Assuming type I error probability α = 0.05 and power of 80%, and effect size of 0.2 G*power calculated that 32 participants would need to be recruited.

To account for potential drop out and balanced randomization, we will aim to recruit 40 participants.

Participants will be recruited through the use of posters around Sheffield Hallam University and the University of Leeds, through emails to staff and students, and contacts at surrounding universities. Potentially eligible participants will be identified through the use of a recruitment questionnaire before being invited to a screening visit for full consideration for the study. All participants will provide written informed consent before participating.

A linear mixed model analysis will be used to assess the effect of kefir on outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-70 years old
* Suffer with poor sleep (measured using the PIttsburg Sleep Quality Index with a score > 5)
* BMI in range of 25-35 kg/m2
* Willingness to consume each study drink daily for 4 weeks and attend the laboratory on 4 separate occasions
* For women: Medication in the form of contraception or HRT providing these have not been modified 3 months prior to the first study day

Exclusion Criteria:

* Intolerance or allergy to milk-based products
* Pregnancy/breastfeeding
* Insufficient English language skills to complete all study questionnaires and perform the cognitive tests
* Gastrointestinal disorders
* Inability to attend the laboratory due to travel/mobility difficulties

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
LDL Cholesterol | 4-weeks
  A blood sample via venepuncture will be taken at baseline and again after 4-weeks of daily consumption of the intervention or control for the assessment of LDL cholesterol. Blood samples will be obtained in a fasted state.
Gut microbiome | 4-weeks
  A stool sample will be collected from participants at baseline and after 4 weeks daily consumption of the intervention and control drink. The composition of the microbiome in stool will be measured by 16s rRNA sequencing.
Sleep quality and duration | 4-weeks
  Sleep quality and duration will be measured objectively and subjectively. For subjective measures, the Pittsburg Sleep Quality Index will be used to assess participant's sleep habits. The tool comprises of 7 sub-components and 18 items, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction. In addition, the Epworth Sleepiness Scale. The Epworth sleepiness scale results range from 0 to 24.
  Participants will also wear a Fitbit Charge 2 watch to track their sleep. Sleep measures will be obtained during the 7-day run in and final week of each study intervention for a total of 4 questionnaires to be completed by each participant and 4 week of objective sleep data.

SECONDARY OUTCOMES:
Blood samples | 4-weeks
  Serum or plasma samples will be obtained via venepuncture for the measurement of insulin, fasting blood glucose, lipids (LDL, HDL), triglycerides, iCAM, vCAM, CRP, and IL-6. All measurements will be taken in a fasted state at each intervention day.
Cognitive function | 4 weeks
  A cognitive test battery consisting of 3 cognitive tests will be used to investigate the effect of the intervention or control on cognitive function. Participants mood will also be assessed using the Positive and Negative Affect Schedule (PANAS) questionnaire that asks participants to rate a series of adjectives describing both positive and negative emotions.
Blood pressure | 4 week
  Blood pressure (systolic blood pressure, diastolic blood pressure and heart rate) will be measured in triplicate using a Vicorder after the paritipcant has rested for 15 minutes upon arrival to the lab. All measurements will be taken in a fasted state.
Pulse Wave Analysis | 4 week
  Carotid to femoral Pulse Wave Velocity (PWV) and Augmentation Index (Aix) will be measured using a Vicorder.
Saliva IgG | 4 week
  Participants will be asked to provide a saliva sample after a 10 minute mouth rinse with water. Saliva samples will be analysed for IgA using ELISA.

OTHER OUTCOMES:
Small intestine bacteria composition | From ingestion of capsules to their excretion
  A subsample of participants will be instructed to ingest SIMBA capsules. Upon retrieval, the capsules will be analysed for the composition of microbiome in capsule fluid by 16s rRNA sequencing and the composition of metabolome in capsule fluid by NMR metabolomics. Capsules will be ingested at baseline and at 4-week time frame in each arm.
Dietary Patterns | 4 days
  During the course of the study, participants will be asked to maintain their normal dietary habits. Participants are asked to record their food and drink consumption for 4-days. This food record will be obtained 4-day prior to each intervention arm and 4-day prior to finishing each intervention arm.
Additional questionnaires | 4-weeks
  The Gastrointestinal Symptom questionnaire comprises 15 items in 5 sections: abdominal pain, reflux, indigestion, diarrhea and constipation. Questionnaire responses will be collected at baseline and after 4 week of ingestion of each study drink.
  In addition, a palatability questionnaire (Visual analogue scale) will be given to the participants at the end of each arm.
Body composition | 4 week
  Height and weight will be measured at each study visit for the purpose of BMI calculation.
  In addition Bioelectrical impedance analysis (BIA) will be used to measure fat-free mass, total body water, percent fat, body cell mass, intracellular water, and extracellular water.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lynn, PhD, Principal Investigator — Sheffield Hallam University
Locations (2):
- United Kingdom (2):
  - University of Leeds, Leeds, West Yorkshire
  - College of Health, Wellbeing and Life Sciences, Sheffield

IPD SHARING:
Plan to Share IPD: No